CLINICAL TRIAL: NCT03144557
Title: Efficacy of an Education Protocol in the Correction of Inhalation Techniques in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of an Education Protocol in the Correction of Inhalation Techniques in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3064
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: COPD; Education
Keywords: Education; COPD; Inhalation Devices
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Education protocol to correct inhalation technique
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Education protocol included 4 individual sessions of verbal and graphic instructions to correct inhalation technique in patients with COPD

SUMMARY:
This study evaluates the implementation of an education protocol and its impact on the correct inhalation technique in COPD patients presenting errors or mistakes. There will be 4 sessions, in each one the inhalation technique will be evaluated using a checklist of steps. Whenever errors are found, the correct use of each device will be educated through verbal explanation and written material will be delivered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD diagnosed by spirometry (presence of a postbronchodilator FEV1 / FVC ratio <0.7)
* Over 40 years old
* Use any of the following devices: metered dose inhaler, HandiHaler, Turbuhaler, Diskus, Aerolizer
* Have at least one error in the inhalation technique
* Signature of informed consent.

Exclusion Criteria:

* Artificial airway
* Cognitive impairment noted in the medical history
* Hearing loss that complicates the compression of simple orders
* Bilateral amaurosis
* Functional dependence for the use of inhalers
* Presence of abnormal movements in the upper limbs that interfere and / or impede the correct use of the devices

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in the inhalation technique | Baseline and every session (48-72 hours)
  If the patient that presented errors or mistakes corrected inhalation technique

SECONDARY OUTCOMES:
Type of error | Baseline
  Frequent errors in inhalation technique using different inhaler devices
Inhalation device | Baseline
  Inhaler that presents the greatest number of mistakes
Patient's characteristics | Baseline
  Characteristics of the patients who do not perform the inhalation technique correctly and those who, despite having completed the education protocol, continue to perform it incorrectly

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Gracia, PT-RT, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molimard M, Raherison C, Lignot S, Balestra A, Lamarque S, Chartier A, Droz-Perroteau C, Lassalle R, Moore N, Girodet PO. Chronic obstructive pulmonary disease exacerbation and inhaler device handling: real-life assessment of 2935 patients. Eur Respir J. 2017 Feb 15;49(2):1601794. doi: 10.1183/13993003.01794-2016. Print 2017 Feb. PMID 28182569
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Hess DR, Kallstrom TJ, Mottram CD, Myers TR, Sorenson HM, Vines DL; American Association for Respiratory Care. Care of the ventilator circuit and its relation to ventilator-associated pneumonia. Respir Care. 2003 Sep;48(9):869-79. PMID 14513820
- [Background] Brocklebank D, Ram F, Wright J, Barry P, Cates C, Davies L, Douglas G, Muers M, Smith D, White J. Comparison of the effectiveness of inhaler devices in asthma and chronic obstructive airways disease: a systematic review of the literature. Health Technol Assess. 2001;5(26):1-149. doi: 10.3310/hta5260. PMID 11701099
- [Background] Rootmensen GN, van Keimpema AR, Jansen HM, de Haan RJ. Predictors of incorrect inhalation technique in patients with asthma or COPD: a study using a validated videotaped scoring method. J Aerosol Med Pulm Drug Deliv. 2010 Oct;23(5):323-8. doi: 10.1089/jamp.2009.0785. PMID 20804428
- [Background] Hesselink AE, Penninx BW, Wijnhoven HA, Kriegsman DM, van Eijk JT. Determinants of an incorrect inhalation technique in patients with asthma or COPD. Scand J Prim Health Care. 2001 Dec;19(4):255-60. doi: 10.1080/02813430152706792. PMID 11822651
- [Background] Goodman DE, Israel E, Rosenberg M, Johnston R, Weiss ST, Drazen JM. The influence of age, diagnosis, and gender on proper use of metered-dose inhalers. Am J Respir Crit Care Med. 1994 Nov;150(5 Pt 1):1256-61. doi: 10.1164/ajrccm.150.5.7952549.
- [Background] van Beerendonk I, Mesters I, Mudde AN, Tan TD. Assessment of the inhalation technique in outpatients with asthma or chronic obstructive pulmonary disease using a metered-dose inhaler or dry powder device. J Asthma. 1998;35(3):273-9. doi: 10.3109/02770909809068218. PMID 9661680
- [Background] Jarvis S, Ind PW, Shiner RJ. Inhaled therapy in elderly COPD patients; time for re-evaluation? Age Ageing. 2007 Mar;36(2):213-8. doi: 10.1093/ageing/afl174. Epub 2007 Jan 31. PMID 17267450
- [Background] Harvey J, Williams JG. Randomised cross-over comparison of five inhaler systems for bronchodilator therapy. Br J Clin Pract. 1992 Winter;46(4):249-51. PMID 1290733
- [Background] van der Palen J, Klein JJ, Kerkhoff AH, van Herwaarden CL. Evaluation of the effectiveness of four different inhalers in patients with chronic obstructive pulmonary disease. Thorax. 1995 Nov;50(11):1183-7. doi: 10.1136/thx.50.11.1183. PMID 8553275
- [Background] Yawn BP, Colice GL, Hodder R. Practical aspects of inhaler use in the management of chronic obstructive pulmonary disease in the primary care setting. Int J Chron Obstruct Pulmon Dis. 2012;7:495-502. doi: 10.2147/COPD.S32674. Epub 2012 Jul 25. PMID 22888221
- [Background] National Clinical Guideline Centre (UK). Chronic Kidney Disease (Partial Update): Early Identification and Management of Chronic Kidney Disease in Adults in Primary and Secondary Care. London: National Institute for Health and Care Excellence (UK); 2014 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK248058/ PMID 25340245
- [Background] Area de asma de SEPAR; Area de enfermeria de SEPAR; Departamento de asma ALAT. [SEPAR-ALAT consensus for inhaled therapies]. Arch Bronconeumol. 2013 Jun;49 Suppl 1:2-14. No abstract available. Spanish. PMID 23967487
- [Background] Myers TR. The science guiding selection of an aerosol delivery device. Respir Care. 2013 Nov;58(11):1963-73. doi: 10.4187/respcare.02812. PMID 24155355
- [Background] Capstick TG, Clifton IJ. Inhaler technique and training in people with chronic obstructive pulmonary disease and asthma. Expert Rev Respir Med. 2012 Feb;6(1):91-101; quiz 102-3. doi: 10.1586/ers.11.89. PMID 22283582
- [Background] Hendeles L, Colice GL, Meyer RJ. Withdrawal of albuterol inhalers containing chlorofluorocarbon propellants. N Engl J Med. 2007 Mar 29;356(13):1344-51. doi: 10.1056/NEJMra050380. No abstract available. PMID 17392304
- [Background] Giner J, Basualdo LV, Casan P, Hernandez C, Macian V, Martinez I, Mengibar A. [Guideline for the use of inhaled drugs. The Working Group of SEPAR: the Nursing Area of the Sociedad Espanola de Neumologia y Cirugia Toracica]. Arch Bronconeumol. 2000 Jan;36(1):34-43. doi: 10.1016/s0300-2896(15)30231-3. No abstract available. Spanish. PMID 10726183
- [Background] Pinto Pereira L, Clement Y, Simeon D. Educational intervention for correct pressurised metered dose inhaler technique in Trinidadian patients with asthma. Patient Educ Couns. 2001 Jan;42(1):91-7. doi: 10.1016/s0738-3991(00)00090-2. PMID 11080609
- [Background] Rau JL. Practical problems with aerosol therapy in COPD. Respir Care. 2006 Feb;51(2):158-72. PMID 16441960
- [Background] van der Palen J, Klein JJ, van Herwaarden CL, Zielhuis GA, Seydel ER. Multiple inhalers confuse asthma patients. Eur Respir J. 1999 Nov;14(5):1034-7. doi: 10.1183/09031936.99.14510349. PMID 10596686
- [Background] McDonald VM, Higgins I, Simpson JL, Gibson PG. The importance of clinical management problems in older people with COPD and asthma: do patients and physicians agree? Prim Care Respir J. 2011 Dec;20(4):389-95. doi: 10.4104/pcrj.2011.00025. PMID 21448550
- [Background] Geller DE. Comparing clinical features of the nebulizer, metered-dose inhaler, and dry powder inhaler. Respir Care. 2005 Oct;50(10):1313-21; discussion 1321-2. PMID 16185367
- [Background] Melani AS, Bracci LS, Rossi M. Reduced Peak Inspiratory Effort through the Diskus((R)) and the Turbuhaler((R)) due to Mishandling is Common in Clinical Practice. Clin Drug Investig. 2005;25(8):543-9. doi: 10.2165/00044011-200525080-00007. PMID 17532698
- [Background] Georges CA, Bolton LB, Bennett C. Functional health literacy: an issue in African-American and other ethnic and racial communities. J Natl Black Nurses Assoc. 2004 Jul;15(1):1-4. PMID 15712814
- [Background] Fink JB, Rubin BK. Problems with inhaler use: a call for improved clinician and patient education. Respir Care. 2005 Oct;50(10):1360-74; discussion 1374-5. PMID 16185371
- [Background] Melani AS, Bonavia M, Cilenti V, Cinti C, Lodi M, Martucci P, Serra M, Scichilone N, Sestini P, Aliani M, Neri M; Gruppo Educazionale Associazione Italiana Pneumologi Ospedalieri. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun;105(6):930-8. doi: 10.1016/j.rmed.2011.01.005. Epub 2011 Mar 2. PMID 21367593
- [Background] Inhaler Error Steering Committee; Price D, Bosnic-Anticevich S, Briggs A, Chrystyn H, Rand C, Scheuch G, Bousquet J. Inhaler competence in asthma: common errors, barriers to use and recommended solutions. Respir Med. 2013 Jan;107(1):37-46. doi: 10.1016/j.rmed.2012.09.017. Epub 2012 Oct 23. PMID 23098685
- [Background] Dolovich MB, Ahrens RC, Hess DR, Anderson P, Dhand R, Rau JL, Smaldone GC, Guyatt G; American College of Chest Physicians; American College of Asthma, Allergy, and Immunology. Device selection and outcomes of aerosol therapy: Evidence-based guidelines: American College of Chest Physicians/American College of Asthma, Allergy, and Immunology. Chest. 2005 Jan;127(1):335-71. doi: 10.1378/chest.127.1.335. PMID 15654001
- [Background] Wright J, Brocklebank D, Ram F. Inhaler devices for the treatment of asthma and chronic obstructive airways disease (COPD). Qual Saf Health Care. 2002 Dec;11(4):376-82. doi: 10.1136/qhc.11.4.376. PMID 12468702
- [Background] Virchow JC, Crompton GK, Dal Negro R, Pedersen S, Magnan A, Seidenberg J, Barnes PJ. Importance of inhaler devices in the management of airway disease. Respir Med. 2008 Jan;102(1):10-9. doi: 10.1016/j.rmed.2007.07.031. Epub 2007 Oct 17. PMID 17923402